CLINICAL TRIAL: NCT01435460
Title: A Clinical Safety and Efficacy Evaluation of Alrex® (Loteprednol Etabonate Ophthalmic Suspension, 0.2%) Versus Patanol (Olopatadine Hydrochloride Ophthalmic Solution, 0.1%) in the Treatment of Seasonal Allergic Conjunctivitis (SAC)
Brief Title: Alrex® Versus Patanol in the Treatment of Seasonal Allergic Conjunctivitis(SAC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 634
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Seasonal Allergic Conjunctivitis
Keywords: ocular allergy
MeSH Terms: interventions — Loteprednol Etabonate; Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alrex (Experimental): Ophthalmic formulation containing the active ingredient loteprednol etabonate, 0.2%
  Interventions: Drug: Loteprednol etabonate 0.2%
- Patanol (Active Comparator): Ophthalmic solution containing olopatadine, 0.1%
  Interventions: Drug: Olopatadine 0.1%

INTERVENTIONS:
Drug: Loteprednol etabonate 0.2% — 1 drop of Alrex 4 times daily (QID) in both eyes at approximately 4 hour intervals for 2 weeks.
  Other Names: Alrex
  Arms: Alrex
Drug: Olopatadine 0.1% — 1 drop of Patanol 2 times daily (BID)at intervals of 6-8 hours or more for 2 weeks.
  Other Names: Patanol
  Arms: Patanol

SUMMARY:
This study is to evaluate the safety and efficacy of Alrex (LE ophthalmic suspension, 0.2%) versus Patanol (olopatadine hydrochloride ophthalmic solution, 0.1%) in the temporary relief of the signs and symptoms of Seasonal Allergic Conjunctivitis (SAC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are diagnosed with acute SAC and experience at least grade 4 ocular itching and at least grade 2 bulbar conjunctival injection (redness) in each eye due to seasonal allergy at Visit 1.

Exclusion Criteria:

* Subjects who have a known hypersensitivity to the study medications or their components or contraindications to ocular corticosteroids.
* Subjects who use any of the disallowed medications throughout the duration of the study and during the period indicated prior to Visit 1.
* Subjects who have intraocular pressure (IOP) greater than 21 mm Hg in either eye or any type of glaucoma.
* Subjects who have a history of any severe/serious ocular pathology or medical condition that could result in the subject's inability to complete the study or affect the subject's safety or trial parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Chu, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Singapore, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Gong L, Sun X, Qu J, Wang L, Zhang M, Zhang H, Wang L, Gu Y, Elion-Mboussa A, Roy L, Zhu B. Loteprednol etabonate suspension 0.2% administered QID compared with olopatadine solution 0.1% administered BID in the treatment of seasonal allergic conjunctivitis: a multicenter, randomized, investigator-masked, parallel group study in Chinese patients. Clin Ther. 2012 Jun;34(6):1259-1272.e1. doi: 10.1016/j.clinthera.2012.04.024. Epub 2012 May 23. PMID 22627057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three hundred participants were enrolled in the study. First participant was enrolled 08/03/2010, last participant exited on 04/26/2011. This study was conducted at 7 sites in China.
Pre-assignment Details: Three hundred participants were randomized into two groups, 151 to be treated with Alrex and 149 to be treated with Patanol.
Period: Overall Study
Arm/Group | Alrex | Patanol
Started | 151 | 149
Completed | 140 | 143
Not Completed | 11 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Did not meet eligibility criteria | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alrex | Patanol | Total
Number analyzed (Participants) | 151 | 149 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 40.5 (14.01) | 40.6 (12.85) | 40.6 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 103 | 202
  Male | 52 | 46 | 98
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 151 | 149 | 300

OUTCOME MEASURES:

1. Primary Outcome: Bulbar Conjunctival Injection
Description: Bulbar conjunctival injection (sign) evaluated using a grading scale from 0-3: where 0 = Absent and 3 = Severe
Time Frame: Change from baseline to day 15 (visit 3)
Population: Participants analyzed from the per protocol (PP) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alrex | Patanol
Number analyzed (Participants) | 138 | 142
units on a scale | -1.91 (0.521) | -1.71 (0.585)

2. Primary Outcome: Ocular Itching
Description: Ocular itching (symptom) evaluated using a grading scale from 0-4 where 0 = Absent and 4 = Severe
Time Frame: Change from baseline to day 15 (visit 3)
Population: Participants analyzed from the per protocol (PP) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alrex | Patanol
Number analyzed (Participants) | 138 | 142
units on a scale | -3.74 (0.469) | -3.28 (0.908)

3. Secondary Outcome: Bulbar Conjunctival Injection
Description: Bulbar conjunctival injection (sign) evaluated using a grading scale from 0-3: where 0 = Absent and 3 = Severe
Time Frame: Change from baseline to day 8 (visit 2)
Population: Participants analyzed from the per protocol (PP) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alrex | Patanol
Number analyzed (Participants) | 140 | 141
units on a scale | -1.36 (0.569) | -1.18 (0.610)

4. Secondary Outcome: Ocular Itching
Description: Ocular itching (symptom) evaluated using a grading scale from 0-4 where 0 = Absent and 4 = Severe
Time Frame: Change from baseline to day 8 (visit 2)
Population: Participants analyzed from the per protocol (PP) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alrex | Patanol
Number analyzed (Participants) | 140 | 141
units on a scale | -2.46 (0.876) | -2.02 (0.851)

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Alrex | Patanol
Serious Adverse Events (participants affected / at risk) | 1/151 | 0/149
Other Adverse Events (participants affected / at risk) | 0/151 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alrex (N=151) | Patanol (N=149)
Deviated Septum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s)after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.